CLINICAL TRIAL: NCT01643850
Title: A Phase II Randomized, Double -Blind, Placebo Controlled Study to Assess Safety, Tolerability and Effect on Tumor Size of MCS110 in Patients With Pigmented Villonodular Synovitis (PVNS)
Brief Title: MCS110 in Patients With Pigmented Villonodular Synovitis (PVNS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMCS110X2201; 2011-002951-32 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-07-18 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Pigmented Villonodular Synovitis; PVNS; Giant Cell Tumor of the Tendon Sheath; GCCTS; Tenosynovial Giant Cell Tumor Localized or Diffused Type; GCTS
Keywords: Pigmented Villonodular Synovitis; PVNS; Giant cell tumor of the tendon sheath; GCCTS; Tenosynovial giant cell tumor (localized or diffused type); GCTS; MCS110
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- MCS110 (Experimental): Participants will receive a single dose of 10mg/kg on day 1 administered by regular infusion.
  Interventions: Drug: MCS110
- Placebo (Placebo Comparator): Part A: single-dose placebo to match MCS110 (10 mg/kg, 1 h i.v. infusion) Part B: single dose placebo to match MCS110 (10 mg/kg, 1 h i.v. infusion administered i.v. at Day 1, followed by 6 doses of placebo to match MCS110 (10 mg/kg)
  Interventions: Drug: Placebo
- MCS110 3 mg/kg (Experimental): Part C: MCS110 3 mg/kg (i.v. infusion)
  Interventions: Drug: MCS110
- MCS110 5 mg/kg (Experimental): Part C: MCS110 5 mg/kg (i.v. infusion)
  Interventions: Drug: MCS110
- MCS110 10 mg/kg (Experimental): Part C: MCS110 10 mg/kg (i.v. infusion)
  Interventions: Drug: MCS110
- MCS110 3 mg/kg & MCS110 10mg/kg (Experimental): Part C: MCS110 3 mg/kg (i.v. infusion) & MCS110 10 mg/kg (i.v. infusion)
  Interventions: Drug: MCS110
- MCS110 5 mg/kg & MCS110 10mg/kg (Experimental): Part C: MCS110 5 mg/kg (i.v. infusion) & MCS110 10 mg/kg (i.v. infusion)
  Interventions: Drug: MCS110

INTERVENTIONS:
Drug: MCS110 — Patients will receive up to 6 doses of MCS110 (3 or 5 or 10mg/kg) administered intravenously once every 4 weeks. Before each dosing, safety will be assessed.
  Other Names: Intravenous infusion of MCS110.
  Arms: MCS110; MCS110 10 mg/kg; MCS110 3 mg/kg; MCS110 3 mg/kg & MCS110 10mg/kg; MCS110 5 mg/kg; MCS110 5 mg/kg & MCS110 10mg/kg
Drug: Placebo — Participants will receive a single dose of NaCl on day 1 through intravenous infusion.
  Other Names: Intravenous infusion of placebo.
  Arms: Placebo

SUMMARY:
This study, designed as a proof of concept study of MCS110 in pigmented villonodular synovitis, assessed the clinical response to MCS110 treatment in Pigmented Villonodular Synovitis (PVNS) patients, after a single or multiple intravenous doses of MCS110, using magnetic resonance imaging to assess tumor volume, and evaluated the pharmacokinetics/pharmacodynamics, safety and tolerability in this population.

ELIGIBILITY:
Inclusion criteria:

* Males and Females aged ≥ 18 years (≥ 12 years in PART C) with PVNS or GCTTS with, at least, one measurable site of disease on MRI.
* Patients expected to get surgery (PART A of study only).
* Vital signs within the ranges: systolic blood pressure 80-150 mmHg , diastolic blood pressure 50-100 mmHg, pulse rate 40-100 bpm, oral body temperature 35.0-37.5°C.
* Patients with normal level of serum ionized calcium and phosphate.
* Women of child-bearing potential must use highly effective contraception during the study and for 84 days after the study drug infusion.

Exclusion criteria:

* Patients with major surgery less than 3 months prior to start study drug or who have still side effects of such therapy.
* Presence of systemic illness precluding definitive surgery or increasing the risk to patients due to potential immunosuppression.
* Use previously of intra-articular treatment within 4 weeks prior dosing.
* Patients with dermal change indicative of lymphedema or phlebolymphedema. disease.
* Patients with elevated troponin T and/or CK levels (> 1.5 x ULN for the laboratory) or with history of myositis, rhabdomyolysis or other myopathic disease.
* Patients receiving immunosuppressive treatment as well as corticosteroids which cannot be discontinued at least 4 weeks before dosing.
* Patients engaged in a resistance exercise training program.
* Patients with pacemakers or any metallic objects as exclusion for MRI
* Patients with concomitant disease know to get influence on bone metabolism
* Patients who have history of drug or alcohol abuse within 12 months prior study dosing.
* Pregnant or nursing (lactating) women.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2018-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (7):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Blay JY, El Sayadi H, Thiesse P, Garret J, Ray-Coquard I. Complete response to imatinib in relapsing pigmented villonodular synovitis/tenosynovial giant cell tumor (PVNS/TGCT). Ann Oncol. 2008 Apr;19(4):821-2. doi: 10.1093/annonc/mdn033. Epub 2008 Feb 21. No abstract available. PMID 18296418
- See also: Ann Oncol. 2008 Apr;19(4):821-2. Epub 2008 Feb 21; Complete response to imatinib in relapsing pigmented villonodular synovitis/tenosynovial giant cell tumor (PVNS/TGCT) — http://www.ncbi.nlm.nih.gov/pubmed/18296418
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven subjects diagnosed with PVNS or GCTTS were evaluated as part of this study. In all, 36 subjects were treated in three parts (Parts A, B and C) of the study, 30 of whom completed the study. At this final analysis, 6 treated subjects had discontinued from the study.
Groups:
- MCS110 10 mg/kg (PART A): Participants received a single dose of 10 mg/kg on Day 1 administered by i.v. infusion
- Placebo (PART A): Participants received single dose placebo by i.v. infusion to match MCS110 10 mg/kg
- MCS110 10 mg/kg (PART B): Participants received multiple monthly doses of MCS110 10 mg/kg. This group also included participants who had received placebo as a 1st dose
- Placebo/10mg/kg (PART B): Participants received single dose placebo to match first dose of MCS110 10 mg/kg and then continued with monthly administration of MCS110 10 mg/kg. fter this first single dose of placebo participants switched to monthly administration of MCS110 10 mg/kg and were added to the MCS110 10 mg/kg (PART B) group, which then increased from 8 to 11 participants. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again
- MCS110 3 mg/kg (Part C): Participants received multiple monthly doses of MCS110 3 mg/kg. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again
- MCS110 5 mg/kg (Part C): Participants received multiple monthly doses of MCS110 5 mg/kg. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again
- MCS110 10 mg/kg (Part C): Participants received multiple monthly doses of MCS110 10 mg/kg. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again
- MCS110 3 mg/kg & MCS110 10mg/kg (Part C): Participants received 3 doses of 3 mg/kg and if not efficacious (≥45% of tumor volume reduction) could switch to 10 mg/kg. This is a subset of participants who started with a dose of 3 mg/kg. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again.
- MCS110 5 mg/kg & MCS110 10mg/kg (PART C): Participants received 3 doses of 5 mg/kg and if not efficacious (≥45% of tumor volume reduction) could switch to 10 mg/kg. This is a subset of participants who started with a dose of 5 mg/kg. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again.
Period: Overall Study
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10mg/kg (PART B) | MCS110 3 mg/kg (Part C) | MCS110 5 mg/kg (Part C) | MCS110 10 mg/kg (Part C) | MCS110 3 mg/kg & MCS110 10mg/kg (Part C) | MCS110 5 mg/kg & MCS110 10mg/kg (PART C)
Started | 5 | 2 | 8 | 3 | 3 | 3 | 4 | 4 | 4
Completed | 5 | 2 | 7 | 3 | 0 | 3 | 3 | 4 | 3
Not Completed | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Administrative Problems | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10mg/kg (PART B) | MCS110 3 mg/kg (Part C) | MCS110 5 mg/kg (Part C) | MCS110 10 mg/kg (Part C) | MCS110 3 mg/kg & MCS110 10mg/kg (Part C) | MCS110 5 mg/kg & MCS110 10mg/kg (PART C) | Total
Number analyzed (Participants) | 5 | 2 | 8 | 3 | 3 | 3 | 4 | 4 | 4 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.4 (8.96) | 30.0 (4.24) | 46.3 (10.14) | 26.7 (11.59) | 45.7 (17.93) | 38.0 (21.66) | 43.8 (13.38) | 46.3 (2.87) | 29.0 (6.06) | 41.3 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 6 | 2 | 1 | 1 | 3 | 2 | 3 | 22
  Male | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 2 | 1 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 4 | 1 | 8 | 2 | 3 | 3 | 3 | 4 | 3 | 31
  Black | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Other | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pigmented Villonodular Synovitis (PVNS) Tumor Size
Description: To assess the efficacy of a single i.v. dose of MCS110 in changing the size of PVNS tumors (as compared to baseline) compared to placebo over 4 weeks evaluated by volume of PVNS tumors by 3-dimensional MRI. This analysis includes all data from patients 4 weeks after receiving the first dose of MCS110 (3, 5 or 10 mg/kg) or placebo and assesses the tumor volume changes at week 4 as compared to baseline. As all parts (Part A, B and C) of the study are assessed after a single dose at week 4 the data set is called "ABC4".
Time Frame: Week 4
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: mm3
Groups:
- Placebo (PART ABC4): Single dose placebo from PART A and B
- MCS110 3 mg/kg (PART ABC4): Single dose MCS110 3 mg/kg. This group included also the subjects who later switch to MCS110 10 mg/kg
- MCS110 5 mg/kg (PART ABC4): Single dose MCS110 5 mg/kg. This group included also the subjects who later switch to MCS110 10 mg/kg.
- MCS110 10 mg/kg (PART ABC4): Single dose MCS110 10 mg/kg
Arm/Group | Placebo (PART ABC4) | MCS110 3 mg/kg (PART ABC4) | MCS110 5 mg/kg (PART ABC4) | MCS110 10 mg/kg (PART ABC4)
Number analyzed (Participants) | 5 | 7 | 7 | 17
mm3 | -4222.8 (6284.56) | -668.5 (18751.44) | -9998.4 (15628.40) | -38002.1 (57314.73)

2. Primary Outcome: Percent Change in Pigmented Villonodular Synovitis (PVNS) Tumor Size
Description: To assess the efficacy of a single i.v. dose of MCS110 in percent change of the PVNS tumor volume at week 4 as compared to baseline and compared to placebo evaluated by volume of PVNS tumors by 3-dimensional MRI. This analysis includes all data from patients who received at least a single dose of MCS110 (3, 5 or 10 mg/kg) or placebo and assesses the tumor volume changes at week 4 as compared to baseline. As all parts (Part A, B and C) of the study are assessed after a single dose at week 4 the data set is called "ABC4".
Time Frame: Week 4
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo (PART ABC4) | MCS110 3 mg/kg (PART ABC4) | MCS110 5 mg/kg (PART ABC4) | MCS110 10 mg/kg (PART ABC4)
Number analyzed (Participants) | 5 | 7 | 7 | 17
Percentage | -7.7 (5.10) | -7.4 (13.21) | -24.8 (23.42) | -32.6 (16.61)
Statistical Analysis 1: Comparison: Placebo (PART ABC4) vs MCS110 3 mg/kg (PART ABC4); Test type: Superiority; p = 0.915, ANCOVA; Mean Difference (Net) = 0.98, 95% CI 2-sided [0.71 to 1.36]
Statistical Analysis 2: Comparison: Placebo (PART ABC4) vs MCS110 5 mg/kg (PART ABC4); Test type: Superiority; p = 0.117, ANCOVA; Median Difference (Net) = 0.78, 95% CI 2-sided [0.57 to 1.07]
Statistical Analysis 3: Comparison: Placebo (PART ABC4) vs MCS110 10 mg/kg (PART ABC4); Test type: Superiority; p = 0.010, ANCOVA; Mean Difference (Net) = 0.69, 95% CI 2-sided [0.52 to 0.91]

3. Primary Outcome: Change in Pigmented Villonodular Synovitis (PVNS) or Giant Cell Tumor of the Tendon Sheath (GCTTS) Tumor Size
Description: Assessment of maximum efficacy (multiple i.v.monthly doses (2 to 6) of 3, 5 or 10 mg/kg MCS110 or 3 & 10 mg/kg or 5 & 10 mg/kg in changing PVNS tumor volume (as compared to baseline) up to 8 weeks post last dose evaluated by MRI. Analysis included data starting from 1st dose of MCS110 in all treatment groups of Parts B and C. Part B patients who received placebo as 1st dose, measurement prior to receiving first dose of MCS110, was used as baseline and assessment time-points were adjusted accordingly. For Part C, participants starting treatment with low dose of MCS110 of 3 or 5 mg/kg could switch to 10 mg/kg after 3 monthly doses, if MCS110 was well tolerated and tumor volume reduction was ≤ 45%. Analysis includes data from patients who received at least 2 doses. The following five groups were assessed: Subjects receiving only 3 mg/kg, only 5 mg/kg or 10 mg/kg and those who switched after 3 doses of 3 mg/kg to 10 mg/kg [3/10 mg/kg] or after 3 doses of 5 mg/kg to 10 mg/kg [5/10 mg/kg]
Time Frame: Up to 8 weeks post last dose
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: mm3
Groups:
- MCS110 3 mg/kg (PART C): Participants received multiple monthly doses of MCS110 3 mg/kg
- MCS110 10 mg/kg (PART BC): Participants received multiple monthly doses of MCS110 10 mg/kg. This included patients who started with single dose placebo, then switched to MCS110 10mg/kg after they switched to MCS110 10mg/kg and had their baseline re-calculated.
- MCS110 5 mg/kg & MCS110 10mg/kg (Part C): Participants received 3 monthly doses of 5 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
Arm/Group | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 10 mg/kg (PART BC) | MCS110 3 mg/kg & MCS110 10mg/kg (Part C) | MCS110 5 mg/kg & MCS110 10mg/kg (Part C)
Number analyzed (Participants) | 7 | 7 | 15 | 4 | 4
mm3 | -2450.3 (2721.24) | -29164.3 (23286.18) | -37015.1 (29297.02) | -42420.1 (63812.69) | -3571.9 (3612.97)

4. Primary Outcome: Percentage Change in Pigmented Villonodular Synovitis (PVNS) or Giant Cell Tumor of the Tendon Sheath (GCTTS) Tumor Size
Description: To assess the maximum efficacy of multiple monthly i.v. doses (2 to 6) of 3, 5 or 10 mg/kg MCS110 or 3 and 10 mg/kg or 5 and 10 mg/kg by percent change in the PVNS tumor volume (as compared to baseline) up to 8 weeks post last dose evaluated by MRI. Subjects starting treatment with a low dose of MCS110 of 3 or 5 mg/kg could switch to 10 mg/kg after 3 monthly doses, if MCS110 was well tolerated and the tumor volume reduction was ≤ 45%. This analysis includes data from all participants who received at least 2 doses of MCS110 and thus includes only patients from Part B and C of the study, thus the data set is called "Part BC". The following five groups were assessed: Subjects receiving only 3 mg/kg, only 5 mg/kg or 10 mg/kg and those who switched after 3 doses of 3 mg/kg to 10 mg/kg [3/10 mg/kg] or after 3 doses of 5 mg/kg to 10 mg/kg [5/10 mg/kg].
Time Frame: Up to 8 weeks post last dose
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- MCS110 3 mg/kg (PART BC): Participants received multiple monthly doses of MCS110 3 mg/kg
- MCS110 5 mg/kg (PART BC): Participants received multiple monthly doses of MCS110 5 mg/kg
- MCS110 3 mg/kg & MCS110 10mg/kg (Part BC): Participants received 3 monthly doses of 3 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
- MCS110 5 mg/kg & MCS110 10mg/kg (Part BC): Participants received 3 monthly doses of 5 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (PART BC) | MCS110 3 mg/kg & MCS110 10mg/kg (Part BC) | MCS110 5 mg/kg & MCS110 10mg/kg (Part BC)
Number analyzed (Participants) | 7 | 7 | 15 | 4 | 4
Percentage | -29.7 (33.73) | -56.3 (20.31) | -55.0 (19.02) | -45.8 (40.11) | -22.6 (16.21)

5. Primary Outcome: Number of Participants With Adverse Events
Description: Overall incidence of Adverse Events
Time Frame: Approximately 2 years
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- MCS110 10 mg/kg (PART A): Participants received a single dose of 10mg/kg on day 1 administered by i.v. infusion.
- Placebo (PART A): Participants received single dose placebo to match MCS110 10mg/kg (i.v. infusion)
- Placebo (PART B): Participants received single dose placebo to match first dose of MCS110 10 mg/kg (i.v. infusion) and then continued with monthly administration of MCS110 10 mg/kg. Subset of MCS110 (Part B)
- MCS110 10 mg/kg (PART C): Participants received multiple monthly doses of MCS110 10 mg/kg. This group includes also participants who had received before 3 monthly doses of 3 or 5 mg/kg and then switched to MCS110 10 mg/kg
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo (PART A) | MCS110 10 mg/kg (PART B) | Placebo (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 10 mg/kg (PART C)
Number analyzed (Participants) | 5 | 2 | 11 | 3 | 7 | 7 | 12
Participants
  AEs of mild severity | 3 | 1 | 11 | 1 | 7 | 6 | 11
  AEs of moderate severity | 1 | 1 | 9 | 2 | 4 | 2 | 5
  AEs of severe severity | 0 | 0 | 4 | 0 | 2 | 1 | 4
  Study drug related AEs | 3 | 1 | 10 | 1 | 7 | 5 | 8
  Serious AEs | 0 | 1 | 2 | 0 | 3 | 1 | 4
  AEs leading to discontinuation | 0 | 0 | 0 | 0 | 2 | 1 | 1

6. Secondary Outcome: Pharmacokinetics of MCS110 Area Under the Serum Concentration-time Curve (AUC)
Description: Pharmacokinetic for a single dose of MCS110 for serum concentration -time curve (AUC).
Time Frame: Day 1 (0 - 5 hr), Day 29, Day 85, Day 112, PART B (Day 1: (0 -5 hr), (Day 85: 0 - 5 hr) PART C (Day 1: 0 -5 hr), (Day 85: 0-5 hr)
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: h* ng/mL
Groups:
- Placebo/10 mg kg (PART B): Participants received single dose placebo to match first dose of MCS110 10 mg/kg (i.v. infusion)and then continued with monthly administration of MCS110 10 mg/kg. Participants could receive a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor growth again
- MCS110 3 mg/kg (PART C): Participants received multiple monthly doses of MCS110 3 mg/kg. Participants could receive a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor growth again
- MCS110 mg/kg (PART C): Participants received multiple monthly doses of MCS110 10 mg/kg. Participants could receive a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor growth again
Arm/Group | MCS110 10 mg/kg (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10 mg kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 mg/kg (PART C)
Number analyzed (Participants) | 5 | 8 | 3 | 6 | 7 | 4
h* ng/mL
  Day 1: number analyzed (Participants) | 5 | 8 | 0 | 6 | 7 | 4
  Day 1 | 75632187 (16664282) | 44258092 (6489002) |  | 12900096 (2373049) | 14559871 (7783073) | 44854588 (9743190)
  Day 29: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Day 29 |  |  | 838099 (171148) |  |  |
  Day 85: number analyzed (Participants) | 0 | 8 | 0 | 0 | 1 | 3
  Day 85 |  | 256238447 (140220044) |  |  | 179084.13 (0) | 999719 (278619)
  Day 112: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Day 112 |  |  | 238619590 (63815086) |  |  |

7. Secondary Outcome: Pharmacokinetics of MCS110 Maximum Concentration (Cmax)
Description: Pharmacokinetic characterization of a single dose of MCS110 for maximum serum concentration (Cmax)
Time Frame: as for outcome 6
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MCS110 10 mg/kg (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10 mg kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 mg/kg (PART C)
Number analyzed (Participants) | 5 | 8 | 3 | 6 | 7 | 4
ng/mL
  Day 1: number analyzed (Participants) | 5 | 8 | 0 | 6 | 7 | 3
  Day 1 | 234800 (40598) | 206750 (32745) |  | 66983 (8493) | 85914 (15539) | 214667 (39119)
  Day 29: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Day 29 |  |  | 194667 (36828) |  |  |
  Day 85: number analyzed (Participants) | 0 | 7 | 0 | 0 | 2 | 3
  Day 85 |  | 309429 (54464) |  |  | 97750 (11667) | 255000 (30199)
  Day 112: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
  Day 112 |  |  | 239000 (55154) |  |  |

8. Secondary Outcome: Pharmacokinetics of MCS110 Total Maximum Concentration (Tmax)
Description: Pharmacokinetic characterization of a single dose of MCS110 for time to maximum concentration (Tmax)
Time Frame: as for outcome 6
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hour (h)
Arm/Group | MCS110 10 mg/kg (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10 mg kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 mg/kg (PART C)
Number analyzed (Participants) | 5 | 8 | 3 | 6 | 7 | 4
hour (h)
  Day 1: number analyzed (Participants) | 5 | 8 | 0 | 6 | 7 | 4
  Day 1 | 2.083 [1.083 to 3.083] | 1.192 [1 to 5.05] |  | 3.125 [1.083 to 5.083] | 5 [0 to 5.033] | 4 [1.083 to 5.067]
  Day 29: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 0
  Day 29 |  |  | 1.467 [1 to 1.5] |  |  |
  Day 85: number analyzed (Participants) | 0 | 7 | 0 | 0 | 2 | 3
  Day 85 |  | 1.25 [1 to 5] |  |  | 3.533 [2.033 to 5.033] | 1.233 [1.083 to 5.05]
  Day 112: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
  Day 112 |  |  | 3.1 [1.017 to 5.183] |  |  |

9. Secondary Outcome: Change in Macrophage-colony Stimulating Factor (M-CSF) Plasma Concentrations Over Time
Description: Pharmacokinetic characterization of a single dose of MCS110 for evaluation of macrophage-colony stimulating factor (M-CSF) plasma concentrations over time
Time Frame: Baseline, Day 1, Day 85, Day 169
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Placebo/MCS110 10mg/kg (PART A): Participants received single dose placebo to match MCS110 10 mg/k
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo/MCS110 10mg/kg (PART A) | MCS110 10 mg/kg (PART B) | Placebo/10 mg kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 mg/kg (PART C)
Number analyzed (Participants) | 5 | 2 | 8 | 3 | 6 | 7 | 4
pg/mL
  Baseline: number analyzed (Participants) | 5 | 2 | 7 | 3 | 6 | 5 | 3
  Baseline | 4694.0 (1375.40) | 4940.0 (650.54) | 5767.1 (1159.12) | 5056.7 (1769.67) | 4778.3 (2078.12) | 5420.0 (3126.20) | 3360.0 (747.46)
  Day 1: number analyzed (Participants) | 4 | 2 | 8 | 3 | 6 | 7 | 3
  Day 1 | 4762.5 (2256.34) | 5060.0 (0) | 6405.0 (4103.80) | 4916.7 (545.19) | 4688.3 (1506.46) | 5281.4 (2687.57) | 4423.3 (1134.43)
  Day 85: number analyzed (Participants) | 4 | 2 | 7 | 3 | 1 | 2 | 3
  Day 85 | 1697500.0 (646445.41) | 4235.0 (544.47) | 4238571.4 (1446575.60) | 4526666.7 (1127578.53) | 4750000.0 (0) | 4060000.0 (0) | 4580000.0 (575065.21)
  Day 169: number analyzed (Participants) | 4 | 2 | 8 | 3 | 1 | 1 | 3
  Day 169 | 173750.0 (103345.30) | 469.0 (1357.65) | 5668750.0 (1928829.68) | 5360000.0 (1173797.26) | 2290000.0 (0) | 4090000.0 (0) | 5480000.0 (1225724.28)

10. Secondary Outcome: Change in Serum C-terminal Type 1 Collagen Peptide Concentrations (CTX-I).
Description: Pharmacodynamic characterization of a single dose of MCS110 by measuring C-terminal telopeptide of Type 1 Collagen peptide (CTX-I), a biomarker of bone resorption. Data measured in participants from three arms: participants from Part A, B and C who received a single dose of 10 mg/kg and had assessment at week 4 (Part ABC4); participants from Part A and B who received placebo ; and participants from Part B and C who received multiple monthly doses of MCS110 (10 mg/kg.) Serum CTX-I data were generated in Part A and Part B. In Part C, samples were collected for serum bone CTX-I analysis. The analysis was not performed, as enough information on compound mode of action was obtained using creatine kinase (CK) and monocytes (hematology) data. Only data from 10mg/kg (single and multiple doses) are available.
Time Frame: Baseline, Week 4, Week 24, Week 104
Population: Pharmacodynamic analysis
Measure: Median (Full Range); unit: ng/mL
Groups:
- MCS110 10 mg/kg (PART ABC4): Participants received a single dose of MCS110 10 mg/kg
- Placebo (PARTS A and B): PART A: Participants received single dose placebo to match MCS110 10mg/kg (i.v. infusion). PART B: Participants received single dose placebo to match first dose of MCS110 10 mg/kg (i.v. infusion) and then continued with monthly administration of MCS110 10 mg/kg.
Arm/Group | MCS110 10 mg/kg (PART ABC4) | Placebo (PARTS A and B) | MCS110 10 mg/kg (PART BC)
Number analyzed (Participants) | 17 | 5 | 17
ng/mL
  Baseline: number analyzed (Participants) | 12 | 5 | 10
  Baseline | 0.3 [0.2 to 0.5] | 0.5 [0.4 to 1.0] | 0.4 [0.2 to 0.6]
  Week 4: number analyzed (Participants) | 11 | 5 | 10
  Week 4 | 0.1 [0.0 to 0.1] | 0.6 [0.2 to 0.8] | 0.1 [0.0 to 0.2]
  Week 24: number analyzed (Participants) | 0 | 0 | 8
  Week 24 |  |  | 0.1 [0.0 to 0.2]
  Week 104: number analyzed (Participants) | 0 | 0 | 5
  Week 104 |  |  | 0.3 [0.2 to 0.8]

11. Secondary Outcome: Number of Participants With Negative Anti-MCS110 Antibody
Description: To assess the immunogenicity of MCS110 in serum anti-MCS110 antibody concentrations
Time Frame: Baseline, throughout the study up to Day 505
Population: Safety analysis set
Measure: Number; unit: Number of Participants
Groups:
- MCS110 10 mg/kg (PART A): Participants received a single dose of 10mg/kg on day 1 administered by regular infusion.
- Placebo (PART A): Participants received single dose placebo to match MCS110 10 mg/kg
- Placebo (PART B): Participants received single dose placebo to match first dose of MCS110 10 mg/kg (i.v. infusion) and then continued with monthly administration of MCS110 10 mg/kg
- MCS110 5 mg/kg (Part C): Participants received multiple monthly doses of MCS110 5 mg/kg
- MCS110 10 mg/kg (Part C): Participants received multiple monthly doses of MCS110 10 mg/kg
- MCS110 5 mg/kg & MCS110 10mg/kg (PART C): Participants received 3 doses of 5 mg/kg and if not efficacious (≥45% of tumor volume reduction) could switch to 10 mg/kg. This is a subset of patients who started with a dose of 5 mg/kg
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo (PART A) | MCS110 10 mg/kg (PART B) | Placebo (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (Part C) | MCS110 10 mg/kg (Part C) | MCS110 3 mg/kg & MCS110 10mg/kg (Part C) | MCS110 5 mg/kg & MCS110 10mg/kg (PART C)
Number analyzed (Participants) | 5 | 2 | 8 | 3 | 3 | 4 | 4 | 4 | 4
Number of Participants
  Baseline: number analyzed (Participants) | 5 | 1 | 8 | 3 | 3 | 3 | 4 | 4 | 4
  Baseline | 5 | 1 | 8 | 3 | 3 | 3 | 3 | 4 | 4
  Day 29: number analyzed (Participants) | 4 | 2 | 8 | 3 | 2 | 4 | 4 | 4 | 3
  Day 29 | 4 | 2 | 8 | 3 | 2 | 4 | 4 | 4 | 3
  Day 85: number analyzed (Participants) | 4 | 2 | 7 | 3 | 1 | 3 | 4 | 3 | 4
  Day 85 | 3 | 2 | 7 | 3 | 1 | 3 | 3 | 3 | 4
  Day 127: number analyzed (Participants) | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 127 | 3 | 1 |  |  |  |  |  |  |
  Day 169: number analyzed (Participants) | 4 | 2 | 7 | 1 | 1 | 3 | 3 | 3 | 4
  Day 169 | 4 | 2 | 7 | 1 | 1 | 3 | 3 | 3 | 4
  Day 336: number analyzed (Participants) | 0 | 0 | 7 | 0 | 0 | 2 | 0 | 0 | 0
  Day 336 |  |  | 7 |  |  | 2 |  |  |
  Day 393: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 4 | 2
  Day 393 |  |  |  |  | 1 | 2 | 4 | 4 | 2
  Day 505: number analyzed (Participants) | 0 | 0 | 8 | 0 | 3 | 4 | 4 | 3 | 2
  Day 505 |  |  | 6 |  | 1 | 4 | 4 | 3 | 2

12. Secondary Outcome: Assessment of Change From Baseline in Joint Range of Motion for Knee Extension and Flexion
Description: To assess the clinical response of joint range of motion following a single i.v. dose of MCS110 or placebo as compared to baseline 4 weeks post-dose evaluated in participants, who had a knee tumor, which was the majority of participants (75%). The analysis includes all data from patients 4 weeks after receiving the first dose of MCS110 (3, 5 or 10 mg/kg) or placebo. As all parts (Part A, B and C) of the study are assessed after a single dose at week 4 the data set is called "ABC4".
Time Frame: Week 4
Population: Pharmacodynamic Analysis Set
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Placebo (PART ABC4) | MCS110 3 mg/kg (PART ABC4) | MCS110 5 mg/kg (PART ABC4) | MCS110 10 mg/kg (PART ABC4)
Number analyzed (Participants) | 5 | 7 | 7 | 17
Degree
  Knee Extension: number analyzed (Participants) | 4 | 3 | 3 | 9
  Knee Extension | -7.3 (4.99) | -12.3 (13.65) | 1.7 (2.89) | -10.3 (26.69)
  Knee Flexion: number analyzed (Participants) | 4 | 3 | 3 | 9
  Knee Flexion | -2.8 (8.85) | 3.7 (13.5) | 13.7 (19.76) | -15.4 (43.13)

13. Secondary Outcome: Assessment of Change From Baseline in Joint Range of Motion for Knee Extension and Flexion
Description: To assess the clinical response of joint range of motion following multiple dose treatment with MCS110 3, 5, or 10 mg/kg evaluated in participants with knee tumor, which was the majority of participants (75%). The data presented are changes from baseline in degree. Participants, who started treatment with a low dose of MCS110 of 3 or 5 mg/kg could switch to 10 mg/kg after 3 monthly doses, if MCS110 was well tolerated and the tumor volume reduction was ≤ 45%. This analysis includes data from participants with knee tumor who received at least 2 doses of MCS110 and thus includes only patients from Part B and C of the study, thus the data set is called "Part BC". The following five groups were assessed: Subjects receiving only 3 mg/kg, only 5 mg/kg or 10 mg/kg and those who switched after 3 doses of 3 mg/kg to 10 mg/kg [3/10 mg/kg] or after 3 doses of 5 mg/kg to 10 mg/kg [5/10 mg/kg].
Time Frame: Week 24/28, Week 104
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Degree
Groups:
- MCS110 10 mg/kg (Part BC): Participants received multiple monthly doses of MCS110 10 mg/kg
Arm/Group | MCS110 3 mg/kg (Part BC) | MCS110 5 mg/kg (Part BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 7 | 7 | 15 | 4 | 4
Degree
  Week 24/28: Knee extension: number analyzed (Participants) | 1 | 1 | 11 | 1 | 3
  Week 24/28: Knee extension | -10.0 (0.00) | 0.0 (0.0) | -10.5 (21.36) | -26 (0.0) | 1 (1.73)
  Week 24/28:(Knee Flexion): number analyzed (Participants) | 1 | 1 | 11 | 1 | 3
  Week 24/28:(Knee Flexion) | -2.0 (0.00) | 8 (0.00) | 9.9 (8.77) | 8 (0.0) | 53.0 (61.54)
  Week 104:(Knee Extension): number analyzed (Participants) | 0 | 1 | 8 | 1 | 2
  Week 104:(Knee Extension) |  | 0 (0) | -3.5 (6.07) | -28.0 (0.00) | 2.5 (3.54)
  Week 104: (Knee Flexion): number analyzed (Participants) | 0 | 1 | 8 | 1 | 2
  Week 104: (Knee Flexion) |  | -6 (0) | 7.5 (11.56) | 10 (0.00) | 70.0 (70.71)

14. Secondary Outcome: Change From Baseline in Joint Pain Using a Visual Analog Scale (VAS)
Description: Measurement of the participant's pain with a 100 mm visual analog scale (VAS) following treatment with MCS110 3, 5, or 10 mg/kg evaluated. Data presented are changes from baseline in degree. Participants were asked to place a line perpendicular to the VAS line at the point that represented her/his pain intensity. Using a ruler, the score was determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the participants mark, providing a score from 0-100. Analysis includes data from participants with knee tumor who received at least 2 doses of MCS110 and thus includes only patients from Part B and C of the study, thus the data set is called "Part BC". The following five groups were assessed: Subjects receiving only 3 mg/kg, only 5 mg/kg or 10 mg/kg and those who switched after 3 doses of 3 mg/kg to 10 mg/kg [3/10 mg/kg] or after 3 doses of 5 mg/kg to 10 mg/kg [5/10 mg/kg].
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 28, Week 40, Week 48, Week 104
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Groups:
- MCS110 3 mg/kg & MCS110 10 mg/kg (PART BC): Participants received 3 monthly doses of 3 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
- MCS110 5 mg/kg & MCS110 10 mg/kg (PART BC): Participants received 3 monthly doses of 5 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (PART BC) | MCS110 3 mg/kg & MCS110 10 mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10 mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
millimeters (mm)
  Baseline: number analyzed (Participants) | 2 | 3 | 15 | 4 | 4
  Baseline | 32 (4.24) | 9.3 (12.74) | 28.6 (21.82) | 39.3 (28.43) | 51.0 (15.64)
  Week 4: number analyzed (Participants) | 2 | 3 | 15 | 4 | 4
  Week 4 | 22.5 (20.51) | 4 (5.29) | 22.5 (23.87) | 32.0 (24.54) | 48.5 (30.71)
  Week 12: number analyzed (Participants) | 1 | 3 | 13 | 4 | 4
  Week 12 | 20 (0) | 2.7 (3.06) | 13.9 (16.01) | 27.5 (26.51) | 33 (26.72)
  Week 24: number analyzed (Participants) | 1 | 1 | 12 | 3 | 4
  Week 24 | 0 (0) | 0 (0) | 21.4 (22.07) | 8.5 (9.33) | 20.3 (28.51)
  Week 28 | 40 (0) | 10.7 (17.62) | 0 (0) | 0 (0) | 0 (0)
  Week 40: number analyzed (Participants) | 1 | 3 | 3 | 4 | 3
  Week 40 | 31 (0) | 3.7 (5.51) | 31.0 (31.38) | 22 (15.81) | 25.7 (31.56)
  Week 48: number analyzed (Participants) | 3 | 3 | 9 | 0 | 0
  Week 48 | 0 (0) | 0 (0) | 21.0 (0) |  |
  Week 104: number analyzed (Participants) | 3 | 3 | 11 | 4 | 2
  Week 104 | 0 (0) | 16.0 (18.03) | 22.4 (24.23) | 17.8 (13.02) | 25.7 (24.7)

15. Secondary Outcome: Time to Relapse
Description: Time to relapse describes the time frame from baseline when the tumor volume increases again after the treatment with MCS110. To be considered a relapse tumor volume had to increase greater than 50% of the difference between tumor volume at baseline and the lowest tumor volume measured by MRI. In this assessment the Part B and Part C patients were analyzed separately. N/A (not available):Data analysis not performed as sample size was not analyzable as no patient had surgery/relapse.
Time Frame: Up to Week 104
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Days
Groups:
- MCS110 10mg/kg (PART B); MCS110 10 mg/kg (PART C): Participants received multiple monthly doses of MCS110 10 mg/kg
- MCS110 5 mg/kg (PART C): Participants received multiple monthly doses of MCS110 5 mg/k. Participants could have received a 2nd treatment cycle (6 x 10 mg/kg MCS110) if tumor grew again
- MCS110 3/10 mg/kg (PART C): Participants received 3 monthly doses of 3 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses
- MCS110 5/10 mg/kg (PART C): Participants received 3 monthly doses of 5 mg/kg and switched to monthly doses of 10 mg/kg (max 3 doses)
Arm/Group | MCS110 10mg/kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 10 mg/kg (PART C) | MCS110 3/10 mg/kg (PART C) | MCS110 5/10 mg/kg (PART C)
Number analyzed (Participants) | 11 | 3 | 3 | 4 | 4 | 4
Days | 337.0 (108.89) | 454.0 (0) | 477.0 (0) | 296.0 (103.24) | NA (NA) — N/A (not available):Data analysis not performed as sample size was not analyzable as no patient had surgery/relapse. | NA (NA) — N/A (not available):Data analysis not performed as sample size was not analyzable as no patient had surgery/relapse.

16. Secondary Outcome: Time to Surgery
Description: Time to surgery describes the time frame from baseline to the time point when participants had surgical removement of PVNS tumor. This could be either residual tumor after the tumor volume was reduced or surgery due to relapse. In this assessment the Part B and Part C patients were analyzed separately. Not Available (NA): Data analysis not performed as sample size was not analyzable as no patient had surgery.
Time Frame: Up to Week 104
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MCS110 10mg/kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 10 mg/kg (PART C) | MCS110 3/10 mg/kg (PART C) | MCS110 5/10 mg/kg (PART C)
Number analyzed (Participants) | 11 | 3 | 3 | 3 | 4 | 4
Days | 387.0 (116.25) | 0 (0) | 0 (0) | 231.0 (0) | NA (NA) — Not Available (NA): Data analysis not performed as sample size was not analyzable as no patient had surgery | NA (NA) — Not Available (NA): Data analysis not performed as sample size was not analyzable as no patient had surgery

17. Secondary Outcome: Average of Health-Related Quality of Life Questionnaire Score for mHAQ
Description: The mHAQ assesses 20 activities in 8 categories related to daily life, which are rated on a 4-point Likert scale. The mHAQ is calculated as the average of the single scores with the following scoring: without difficulty =0; with some difficulty =1; with much difficulty =2; unable to do =3. Total score is between 0 - 3.0. Values <0.3 are considered normal. Data presented include only participants, who received multiple doses of MCS110.
Time Frame: up to 104 weeks
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Scores on a scale
  Baseline: number analyzed (Participants) | 2 | 3 | 15 | 4 | 4
  Baseline | 0.3 (0.35) | 0.1 (0.22) | 0.3 (0.20) | 0.3 (0.33) | 0.9 (0.52)
  Week 104: number analyzed (Participants) | 0 | 3 | 11 | 4 | 3
  Week 104 |  | 0.1 (0.14) | 0.2 (0.18) | 0.1 (0.19) | 0.3 (0.25)

18. Secondary Outcome: Number of CD14+ Monocytes and Number of CD14 + Monocytes and CD16+ Monocytes
Description: Blood samples were collected for the evaluation of CD14+ monocytes (using FACS) and CD14+ CD16+ monocytes. Based on preliminary analysis, the quality of the samples did not allow meaningful conclusions to be drawn. Thus, in Part B, the monocyte sample collection was discontinued.
Time Frame: Baseline Up to Week 104
Population: Pharmacodynamic analysis set
Measure: Number; unit: Number of Monocytes
Groups:
- MCS110 3 mg/kg (PART C): Participants received multiple monthly doses of MCS110 5 mg/kg
- MCS110 10 mg/kg (PART C): Participants received multiple monthly doses of MCS110 10 mg/kg )
- MCS110 3 mg/kg & MCS110 10mg/kg (PART C): Participants received 3 doses of 3 mg/kg and if not efficacious (≥45% of tumor volume reduction) could switch to 10 mg/kg. This is a subset of patients who started with a dose of 3 mg/kg
Arm/Group | MCS110 10 mg/kg (PART A) | MCS110 10 mg/kg (PART B) | MCS110 3 mg/kg (PART C) | MCS110 5 mg/kg (PART C) | MCS110 10 mg/kg (PART C) | MCS110 3 mg/kg & MCS110 10mg/kg (PART C) | MCS110 5 mg/kg & MCS110 10mg/kg (PART C)
Number analyzed (Participants) | 5 | 8 | 3 | 3 | 4 | 4 | 4
Number of Monocytes | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done. | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done. | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done. | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done | NA — Due to poor quality, high percentage of samples were not analyzed or results did not meet the acceptance criteria. Because of the paucity of CD14+ and CD14+CD16+ monocytes data no meaningful interpretation could be done

19. Secondary Outcome: Change From Baseline Per Treatment for Activities of Daily Living (ADL) in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a patient-reported outcome measurement instrument developed to assess the subject's opinion about their knee and associated problems. The KOOS questionnaire collected data on 5 knee-specific patient-centered outcomes: activities of daily life (ADL), knee related quality of life (QOL), pain and discomfort, sport/recreation, symptoms. The 5 KOOS sub-scales were scored separately on a Likert scale scored from 0 (no problems) to 4 (extreme problems) and scores were transformed to a 0.100 scale with 0 representing extreme knee problems and 100 representing no problems. The 5 dimensions were analyzed independently. Positive changes (i.e. increases in the score) are beneficial. KOOS was assessed in Part B and C only in participants with knee PVNS tumor.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 48, Week 40, Week 72, Week 104 (end of study)
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Baseline-ADL: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Baseline-ADL | 65.4 (3.12) | 69.1 (0.00) | 77.3 (7.87) | 70.6 (0.00) | 71.3 (30.16)
  Week 4-ADL: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Week 4-ADL | 79.4 (20.8) | 91.2 (0.00) | 86.5 (10.37) | 89.7 (0.00) | 76.0 (18.97)
  Week 12-ADL: number analyzed (Participants) | 1 | 1 | 10 | 1 | 3
  Week 12-ADL | 72.1 (0.00) | 97.1 (0.00) | 87.4 (15.10) | 94.1 (0.00) | 76.5 (23.53)
  Week 24-ADL: number analyzed (Participants) | 1 | 1 | 9 | 1 | 1
  Week 24-ADL | 55.9 (0.00) | 0 (0) | 89.6 (10.75) | 79.4 (0) | 73.0 (28.83)
  Week 28-ADL: number analyzed (Participants) | 3 | 3 | 9 | 0 | 0
  Week 28-ADL | 52.9 (0) | 83.8 (0) | 0 (0) |  |
  Week 40- ADL: number analyzed (Participants) | 1 | 1 | 2 | 1 | 2
  Week 40- ADL | 79.4 (0) | 95.6 (0) | 73.5 (29.12) | 89.7 | 89.0 (15.6)
  Week 48-ADL: number analyzed (Participants) | 0 | 0 | 8 | 0 | 0
  Week 48-ADL |  |  | 85.3 (13.50) |  |
  Week 72-ADL: number analyzed (Participants) | 3 | 1 | 10 | 1 | 2
  Week 72-ADL | 48.5 (0) | 88.2 (0) | 78.7 (20.82) | 91.2 (0) | 100 (0)
  Week 104- ADL: number analyzed (Participants) | 0 | 1 | 7 | 1 | 2
  Week 104- ADL |  | 77.9 | 93.5 (7.74) | 97.1 (0) | 87.5 (17.68)

20. Secondary Outcome: Change From Baseline Per Treatment for Knee Related Quality of Life in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a patient-reported outcome measurement instrument developed to assess the subject's opinion about their knee and associated problems. The KOOS questionnaire collected data on 5 knee-specific patient-centered outcomes: activities of daily life (ADL), knee related quality of life, pain and discomfort, sport/recreation, symptoms. The 5 KOOS sub-scales were scored separately on a Likert scale scored from 0 (no problems) to 4 (extreme problems) and scores were transformed to a 0.100 scale with 0 representing extreme knee problems and 100 representing no problems. The 5 dimensions were analyzed independently. Positive changes (i.e. increases in the score) are beneficial. KOOS was assessed in Part B and C only in participants with knee PVNS tumor.
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 48, Week 40, Week 72, Week 104 (end of study)
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Baseline-Knee: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Baseline-Knee | 15.6 (13.26) | 37.5 (0) | 29.5 (23.23) | 50.0 (0) | 40.6 (4.42)
  Week 4-Knee: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Week 4-Knee | 31.3 (17.68) | 56.3 (0) | 43.8 (22.88) | 43.8 (0) | 45.8 (13.01)
  Week 12-Knee: number analyzed (Participants) | 1 | 1 | 10 | 1 | 3
  Week 12-Knee | 37.5 (0) | 56.3 (0) | 54.4 (28.72) | 62.5 (0) | 43.8 (16.54)
  Week 24-Knee: number analyzed (Participants) | 1 | 0 | 9 | 1 | 3
  Week 24-Knee | 43.8 (0) |  | 50.7 (34.30) | 43.8 (0) | 41.7 (21.95)
  Week 28-Knee: number analyzed (Participants) | 1 | 1 | 9 | 1 | 1
  Week 28-Knee | 12.5 (0) | 56.3 (0) | 46.9 (0) | 68.8 (0) | 56.3 (0)
  Week 40- Knee: number analyzed (Participants) | 1 | 1 | 2 | 1 | 2
  Week 40- Knee | 37.5 (0) | 62.5 (0) | 37.5 (0) | 50.0 (0) | 68.8 (8.84)
  Week 48-Knee: number analyzed (Participants) | 0 | 0 | 8 | 0 | 0
  Week 48-Knee |  |  | 48.4 (25.61) |  |
  Week 72-Knee: number analyzed (Participants) | 1 | 1 | 10 | 1 | 1
  Week 72-Knee | 25.0 (0) | 56.3 (0) | 45.0 (26.81) | 68.8 (0) | 68.8 (0)
  Week 104- Knee: number analyzed (Participants) | 0 | 1 | 7 | 1 | 2
  Week 104- Knee |  | 50.0 (0) | 59.8 (21.61) | 68.8 (0) | 62.5 (17.68)

21. Secondary Outcome: Change From Baseline Per Treatment for Pain and Discomfort in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 20
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 48, Week 40, Week 72, Week 104 (end of study)
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Baseline: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Baseline | 54.2 (5.89) | 52.8 (0) | 62.6 (17.50) | 66.7 (0) | 61.1 (23.57)
  Week 4: number analyzed (Participants) | 2 | 1 | 11 | 1 | 2
  Week 4 | 66.7 (19.64) | 75.0 (0) | 73.5 (18.19) | 75.0 (0) | 63.0 (0)
  Week 12: number analyzed (Participants) | 1 | 1 | 10 | 1 | 3
  Week 12 | 55.6 (0) | 80.6 (0) | 75.6 (20.32) | 75.0 (0) | 71.3 (15.80)
  Week 24: number analyzed (Participants) | 1 | 0 | 9 | 1 | 3
  Week 24 | 52.8 (0) |  | 77.5 (21.22) | 61.1 (0) | 69.4 (25.46)
  Week 28: number analyzed (Participants) | 1 | 1 | 2 | 1 | 1
  Week 28 | 55.6 (0) | 69.4 (0) | 70.8 (41.25) | 83.3 (0) | 88.9 (0)
  Week 40: number analyzed (Participants) | 1 | 1 | 2 | 1 | 2
  Week 40 | 58.3 (0) | 77.8 (0) | 56.9 (0) | 80.6 (0) | 79.2 (21.61)
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 0 | 0
  Week 48 |  |  | 71.5 (21.45) |  |
  Week 72: number analyzed (Participants) | 1 | 1 | 10 | 1 | 1
  Week 72 | 47.2 (0) | 66.7 (0) | 62.2 (25.43) | 88.9 (0) | 91.7 (0)
  Week 104: number analyzed (Participants) | 0 | 1 | 7 | 1 | 2
  Week 104 |  | 58.3 (0) | 77.7 (13.12) | 91.7 (0) | 72.2 (27.50)

22. Secondary Outcome: Change From Baseline Per Treatment for Sport/Recreation in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 20
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 48, Week 40, Week 72, Week 104 (end of study)
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Baseline: number analyzed (Participants) | 2 | 1 | 10 | 1 | 2
  Baseline | 35.0 (7.07) | 25.0 (0) | 29.5 (23.15) | 70.0 (0) | 52.5 (31.82)
  Week 4: number analyzed (Participants) | 2 | 1 | 11 | 1 | 3
  Week 4 | 50.0 (21.21) | 70.0 (0) | 40.9 (0) | 100.0 (0) | 48.3 (45.37)
  Week 12: number analyzed (Participants) | 1 | 1 | 10 | 1 | 3
  Week 12 | 45.0 (0) | 85.0 (0) | 58.0 (0) | 85.0 (0) | 45.0 (37.75)
  Week 24: number analyzed (Participants) | 1 | 0 | 9 | 1 | 3
  Week 24 | 30.0 (0) |  | 55.6 (30.66) | 50.0 (0) | 53.3 (37.53)
  Week 28: number analyzed (Participants) | 1 | 1 | 2 | 1 | 1
  Week 28 | 35.0 (0) | 35.0 (0) | 50.0 (70.71) | 95.0 (0) | 95.0 (0)
  Week 40: number analyzed (Participants) | 1 | 1 | 2 | 1 | 2
  Week 40 | 35.0 (0) | 50.0 (0) | 37.5 (53.03) | 90.0 (0) | 80.0 (21.21)
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 0 | 0
  Week 48 |  |  | 48.1 (39.27) |  |
  Week 72: number analyzed (Participants) | 1 | 1 | 10 | 1 | 1
  Week 72 | 30.0 (0) | 40.0 (0) | 40.6 (36.27) | 70.0 (0) | 95.0 (0)
  Week 104: number analyzed (Participants) | 0 | 1 | 7 | 1 | 2
  Week 104 |  | 30.0 (0) | 58.2 (21.54) | 95.0 (0) | 70.0 (35.36)

23. Secondary Outcome: Change From Baseline Per Treatment for Symptoms in the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: as for outcome 20
Time Frame: Baseline, Week 4, Week 12, Week 24, Week 48, Week 40, Week 72, Week 104 (end of study)
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Baseline: number analyzed (Participants) | 2 | 1 | 10 | 1 | 2
  Baseline | 41.1 (12.63) | 50.0 (0) | 50.0 (16.44) | 50.0 (0) | 62.5 (27.78)
  Week 4: number analyzed (Participants) | 2 | 1 | 11 | 1 | 3
  Week 4 | 58.9 (32.83) | 75.0 (0) | 59.4 (16.92) | 57.1 (0) | 57.1 (24.74)
  Week 12: number analyzed (Participants) | 1 | 1 | 10 | 1 | 3
  Week 12 | 71.4 (0) | 78.6 (0) | 69.3 (21.31) | 64.3 (0) | 56.0 (26.33)
  Week 24: number analyzed (Participants) | 1 | 0 | 9 | 1 | 3
  Week 24 | 50.0 (0) |  | 65.9 (25.45) | 67.9 (0) | 67.9 (0)
  Week 28: number analyzed (Participants) | 1 | 1 | 2 | 1 | 1
  Week 28 | 60.7 (0) | 60.7 (0) | 62.5 (53.03) | 75.0 (0) | 89.3 (0)
  Week 40: number analyzed (Participants) | 1 | 1 | 2 | 1 | 2
  Week 40 | 75.0 (0) | 64.3 (0) | 42.9 (60.61) | 78.6 (0) | 73.2 (37.88)
  Week 48: number analyzed (Participants) | 0 | 0 | 8 | 0 | 0
  Week 48 |  |  | 62.1 (24.29) |  |
  Week 72: number analyzed (Participants) | 1 | 1 | 10 | 1 | 1
  Week 72 | 50.0 (0) | 57.1 (0) | 40.6 (28.43) | 78.6 (0) | 85.7 (0)
  Week 104: number analyzed (Participants) | 0 | 1 | 7 | 1 | 2
  Week 104 |  | 53.6 (0) | 67.3 (20.63) | 85.7 (0) | 62.5 (32.83)

24. Secondary Outcome: Change From Baseline Per Treatment Using EuroQol-5 Dimensional (EQ-5D VAS)Visual Analog Scale Quality of Life Questionnaire
Description: The EQ-5D is a standardized measure of health status. The EQ visual analogue scale (EQ VAS)has a range from 0-100: worst possible to perfect health. Data show the absolute change from baseline of EQ5D VAS and at the different visits for participants, who received multiple doses of MCS110. (PART B and PART C).
Time Frame: Week 4, Week 24, up to 104 weeks
Population: Pharmacodynamic analysis set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MCS110 3 mg/kg (PART BC) | MCS110 5 mg/kg (PART BC) | MCS110 10 mg/kg (Part BC) | MCS110 3 mg/kg & MCS110 10mg/kg (PART BC) | MCS110 5 mg/kg & MCS110 10mg/kg (PART BC)
Number analyzed (Participants) | 3 | 3 | 15 | 4 | 4
Score on a scale
  Week 4: number analyzed (Participants) | 2 | 3 | 15 | 4 | 4
  Week 4 | 11.0 (1.41) | 3.7 (5.03) | 0.6 (25.07) | 1.3 (2.50) | 5.5 (10.85)
  Week 24: number analyzed (Participants) | 1 | 1 | 12 | 3 | 4
  Week 24 | -1.0 (0.00) | 10.0 (0.00) | 9.5 (14.04) | 1.0 (8.54) | 9.8 (16.21)
  Up to Week 104: number analyzed (Participants) | 0 | 3 | 11 | 4 | 3
  Up to Week 104 |  | 1.3 (5.51) | 6.9 (13.93) | 7.0 (8.91) | 18.0 (25.63)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events .Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 2 years.
Groups:
- MCS110 10mg/kg (PART B); MCS110 10mg/kg (PART C): MCS110 10 mg/kg (i.v. infusion)
- MCS110 3mg/kg (PART C): MCS110 3 mg/kg (i.v. infusion)
- MCS110 5mg/kg (PART C): MCS110 5 mg/kg (i.v. infusion)
Arm/Group | MCS110 10 mg/kg (PART A) | Placebo (PART A) | MCS110 10mg/kg (PART B) | Placebo/10mg/kg (PART B) | MCS110 3mg/kg (PART C) | MCS110 5mg/kg (PART C) | MCS110 10mg/kg (PART C)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2 | 0/11 | 0/3 | 0/7 | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/2 | 2/11 | 0/3 | 3/7 | 1/7 | 4/12
Other Adverse Events (participants affected / at risk) | 3/5 | 1/2 | 11/11 | 3/3 | 7/7 | 6/7 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110 10 mg/kg (PART A) (N=5) | Placebo (PART A) (N=2) | MCS110 10mg/kg (PART B) (N=11) | Placebo/10mg/kg (PART B) (N=3) | MCS110 3mg/kg (PART C) (N=7) | MCS110 5mg/kg (PART C) (N=7) | MCS110 10mg/kg (PART C) (N=12)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningoencephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCS110 10 mg/kg (PART A) (N=5) | Placebo (PART A) (N=2) | MCS110 10mg/kg (PART B) (N=11) | Placebo/10mg/kg (PART B) (N=3) | MCS110 3mg/kg (PART C) (N=7) | MCS110 5mg/kg (PART C) (N=7) | MCS110 10mg/kg (PART C) (N=12)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dark circles under eyes (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 4 | 0 | 5 | 3 | 4
Periorbital swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 1 | 3 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Administration site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 4 | 0 | 5 | 2 | 2
Infusion site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 2 | 0 | 2 | 3 | 3
Pyrexia (General disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 0
Soft tissue inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 0 | 1 | 2 | 3
Peritonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Antinuclear antibody positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 4 | 0 | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Benign joint neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 0 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 4 | 0 | 2 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 2 | 2 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 1 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT01643850/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT01643850/SAP_001.pdf